CLINICAL TRIAL: NCT04969861
Title: A Phase 2/3, Randomized, Open-label Study to Compare Bempegaldesleukin Combined With Pembrolizumab Versus Pembrolizumab Alone in First-Line Treatment of Patients With Metastatic or Recurrent Head and Neck Squamous-Cell Carcinoma With PD-L1 Expressing Tumors (PROPEL-36)
Brief Title: BEMPEG With Pembrolizumab vs Pembrolizumab Alone in Patients With Metastatic or Recurrent HNSCC (PROPEL-36)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Nektar Therapeutics made the decision to discontinue the bempegaldesleukin program based on three negative studies. SFJ Pharmaceuticals, Inc. and Nektar Therapeutics, in consultation with the study IDMC, have decided to discontinue PROPEL-36.
Sponsor: Nektar Therapeutics (Industry)
Collaborators: SFJ Pharmaceuticals, Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-214-36
Record Dates: First submitted 2021-07-09; First posted 2021-07-21 (Actual); Results first posted 2022-12-15 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-11

CONDITIONS: Metastatic Head and Neck Cancer; Recurrent Head and Neck Cancer
Keywords: Head and Neck Cancer; Head and Neck Squamous-Cell Carcinoma; HNSCC; BEMPEG; Bempegaldesleukin; NKTR-214; Keytruda; Pembrolizumab; PROPEL-36
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — bempegaldesleukin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BEMPEG + Pembrolizumab (Experimental): Bempegaldesleukin plus pembrolizumab every 3 weeks (q3w) for up to 35 cycles (approximately 2 years).
  Interventions: Drug: Bempegaldesleukin; Drug: Pembrolizumab
- Pembrolizumab Monotherapy (Active Comparator): Pembrolizumab monotherapy q3w for up to 35 cycles (approximately 2 years).
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Bempegaldesleukin — Specified dose on specified days
  Arms: BEMPEG + Pembrolizumab
Drug: Pembrolizumab — Pembrolizumab (anti-PD-1) will be dosed as per the pharmacy manual.

SUMMARY:
This is a multicenter, randomized, open-label, Phase 2/3 study that will evaluate the efficacy and safety of bempegaldesleukin (BEMPEG; NKTR-214) combined with pembrolizumab compared with pembrolizumab monotherapy in patients with recurrent or metastatic HNSCC with positive PD-L1 expression (CPS ≥ 1).

ELIGIBILITY:
Inclusion Criteria:

* Provide written, informed consent to participate in the study and follow the study procedures.
* Male or female patients, age 18 years or older at the time of signing the informed consent form (ICF).
* Have histologically or cytologically-confirmed recurrent or metastatic HNSCC that is considered incurable by local therapies.

  * No prior systemic therapy for recurrent or metastatic disease.
  * The eligible primary tumor locations are oropharynx, oral cavity, hypopharynx, and larynx.
  * Patients may not have a primary tumor site of nasopharynx (any histology) and/or unknown primary.
* Have measurable disease based on RECIST 1.1 as determined by the local site Investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Measure Description: GRADE - ECOG PERFORMANCE STATUS

0 - Fully active, able to carry on all pre-disease performance without restriction

1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work

2- Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours

• The tumor must have positive PD-L1 expression (i.e., CPS ≥1)

Exclusion Criteria:

* Has disease that is suitable for local therapy administered with curative intent.
* Has progressive disease within 6 months of completion of curatively intended systemic treatment for locoregionally advanced HNSCC.
* Has had radiation therapy (or other non-systemic therapy) within 2 weeks prior to initiation of study drug
* Has a life expectancy of less than 3 months and/or has rapidly progressing disease (e.g., tumor bleeding, uncontrolled tumor pain) as determined by the Investigator.
* Has a known additional malignancy that is progressing or has required active treatment within 5 years prior to the first dose of study drug
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy
* Use of an investigational agent or an investigational device within 28 days before the first dose of study drug.
* Prior treatment with an anti PD-1, anti PD-L1, anti-PD-L2, or anti CTLA-4 antibody, agents that target IL-2 pathway, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.

NOTE: Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (4):
- Nebraska Methodist Hospital, Omaha, Nebraska, United States
- Universitätsklinikum Salzburg, Landeskrankenhaus,, Salzburg, Salzburg Bundesland, Austria
- Attikon University General Hospital, Athens, Attica, Greece
- ASST Degli Spedali Civili di Brescia, Brescia, Lombardy, Italy

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BEMPEG + Pembrolizumab | Pembrolizumab Monotherapy
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Study was terminated in consonance with discontinuation of bempegaldesleukin program. | 1 | 0

BASELINE CHARACTERISTICS:
Population: Following the Sponsor's decision to end the trial, treatment was discontinued after one patient received 2 cycles of BEMPEG + Pembrolizumab
Groups:
- Total: Total of all reporting groups
Arm/Group | BEMPEG + Pembrolizumab | Pembrolizumab Monotherapy | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 1 |  | 1
Age, Continuous [Mean (Full Range); unit: years] | 69 [69 to 69] |  | 69 [69 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  Austria | 0 |  | 0
  Greece | 0 |  | 0
  United States | 1 |  | 1
  Italy | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: Approximately 2 years
Population: Nektar and BMS Study PIVOT-IO-001 did not meet its primary EP of demonstrating an efficacy advantage from addition of BEMPEG to nivolumab in patients with previously untreated inoperable or metastatic melanoma. PIVOT-09 (RCC) and PIVOT-10 (uroth C) studies also reported negative topline results. Based on these 3 large negative studies, Nektar and SFJ in consultation with the study IDMC made the decision to discontinue this trial. At termination, 1 patient was enrolled and treated for 2 cycles.
Arm/Group | BEMPEG + Pembrolizumab | Pembrolizumab Monotherapy
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Objective Response Rate
Description: To compare the objective response rate (ORR) of bempegaldesleukin plus pembrolizumab versus pembrolizumab monotherapy.
Time Frame: Approximately 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Progression-Free Survival
Description: To compare progression-free survival (PFS) of bempegaldesleukin plus pembrolizumab versus pembrolizumab monotherapy.
Time Frame: Approximately 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Time to Deterioration
Description: The time from baseline to a ≥ 10-point decrease with confirmation by the subsequent visit of a ≥ 10-point deterioration from baseline in:
  • Global health status/quality of life assessment based on the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30).
  The EORTC QLQ-C30 is a 30-item questionnaire designed to assess the quality of life of cancer patients. All scale scores are linearly converted to range from 0 to 100. A higher total score indicates a better level of functioning.
  • Pain and Swallowing based on respective multi-item scales of EORTC QLQ head and neck cancer specific module (EORTC QLQ-H&N35).
  EORTC QLQ-H&N35 consists of 7 multi-item scales that assess pain, swallowing, senses, speech, social eating, social contact and sexuality. All scale scores are linearly converted to range from 0 to 100. A higher total score indicates increased severity of symptoms.
Time Frame: Approximately 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Change in Global Health Status/Quality of Life
Description: To compare mean change from baseline in global health status/quality of life scale of EORTC QLQ-C30. The EORTC QLQ-C30 is composed of multi-item scales and single item measures. These include 5 functional scales (physical, role, emotional, cognitive, and social), 3 symptom scales (fatigue, nausea/vomiting, and pain), a global health status/HRQoL scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All scale scores are linearly converted to range from 0 to 100. A higher total score indicates a better level of functioning.
Time Frame: Approximately 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Percentage of Patients With Treatment-Emergent Adverse Events and Serious Adverse Events
Description: Compare the overall safety and tolerability based on assessments of treatment-emergent adverse events and serious adverse events
Time Frame: Screening baseline through end of study, approximately 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 month
Description: There were no SAEs, no mortalities. In total, one Grade 1 AE of cough was reported.
Arm/Group | BEMPEG + Pembrolizumab | Pembrolizumab Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BEMPEG + Pembrolizumab (N=1) | Pembrolizumab Monotherapy (N=0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions to the PI's rights to discuss or publish trial results.

DOCUMENTS (2):
  • Study Protocol (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT04969861/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT04969861/SAP_001.pdf